CLINICAL TRIAL: NCT00208234
Title: The Effects of Xolair (Omalizumab) on Airway Hyperresponsiveness
Brief Title: Effect of Xolair on Airway Hyperresponsiveness
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Creighton University (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Xolair Asthma
Record Dates: First submitted 2005-09-14; First posted 2005-09-21 (Estimated); Last update posted 2011-09-23 (Estimated); Status verified 2011-09

CONDITIONS: Allergic Asthma
Keywords: asthma
MeSH Terms: conditions — Asthma | interventions — Omalizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Placebo Comparator): Placebo
  Interventions: Drug: Placebo for Omalizumab
- 2 (Experimental): Omalizumab
  Interventions: Drug: Omalizumab

INTERVENTIONS:
Drug: Omalizumab — 0.016 mg/kg IgE
  Other Names: Xolair; rHuMAbE25
  Arms: 2
Drug: Placebo for Omalizumab — Placebo
  Arms: Control
Drug: omalizumab — Monoclonal antibody against IgE. 0.016 mg/kg IgE
  Other Names: Xolair; rhumabE25
  Arms: 2

SUMMARY:
The purpose of this study is to determine if Xolair can reduce the abnormal increase in limitation to airflow in patients with asthma in a relatively short time period. Another purpose is to determine if Xolair will decrease the amount of inflammation in the lungs of an asthmatic patient in the same time period.

DETAILED DESCRIPTION:
Xolair, a recombinant humanized monoclonal anti-IgE antibody, has been studied extensively and proven efficacious in the treatment of asthma and other allergic disorders. In moderate to severe allergic asthmatic patients, Xolair reduced asthma exacerbations and improved symptoms. However, there is limited data on the effects of Xolair on airway hyperreactivity, an important component of asthma.

ELIGIBILITY:
Inclusion Criteria:

* Female patients must have a negative urine pregnancy test at Visit 1 and a negative urine pregnancy test at subsequent visits. In addition, female patients must be using a medically acceptable form of birth control.
* History of mild to moderate asthma
* A positive skin prick test to one or more perennial environmental allergens (dog, cat, dermatophagoides farinae, or dermatophagoides pteronyssinus)
* A PC20 value for methacholine < 5 mg/mL
* A PC15 value for hypertonic saline at < 4 minutes
* Capable of faithfully attending regularly scheduled study visits
* Willing to avoid prohibited medications for the periods indicated in the protocol
* A baseline serum IgE level of > 30 IU/mL and < 700 IU/mL

Exclusion Criteria:

* Women of childbearing potential not using a medically acceptable form of birth control, as well as women who are breastfeeding
* Known sensitivity to study drug or class of study drug
* Any sinus, middle ear, oropharyngeal, upper or lower respiratory tract infection that has not resolved at least 2 weeks prior to the screening visit, or for which antibiotic therapy has not been completed at least 2 weeks prior to the screening visit
* Patients with a history of severe anaphylactoid or anaphylactic reactions
* Patients taking beta-adrenergic antagonists in any form
* Patients previously exposed to Xolair
* Patients with a known hypersensitivity to trial drug excipient ingredients or related drugs
* Chronic or intermittent use of inhaled, oral, intranasal, intramuscular, or intravenous corticosteroids, or use of topical corticosteroids other than intermittent use of low potency preparations
* Use of immunosuppressive medications
* History or presence of significant renal, hepatic, neurologic, cardiovascular, hematologic, metabolic, cerebrovascular, respiratory, gastrointestinal, or other significant medical condition, including autoimmune or collagen vascular disorders aside from organ-specific autoimmune disease limited to the thyroid that in the investigator's opinion could interfere with the study or require medical treatment that would interfere with the study

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Estimated)
Dates: Start 2004-01; Primary Completion 2011-09 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
To determine if treatment with omalizumab induces changes in PC20 values to methacholine bronchoprovocation challenges and/or PC15 values to hypertonic saline-induced bronchoprovocation challenges in a time-dependent manner in steroid naive subjects | post treatment

SECONDARY OUTCOMES:
Determine in steroid naive allergic asthma subjects whether omalizumab decreases exhaled NO and sputum eosinophilia, markers of airway inflammation, in time-dependent fashion and to correlate these effects with those measured for airway responsiveness | post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Thomas B Casale, MD, Principal Investigator — Creighton University Medical Center
Locations (1):
- Creighton University Division of Allergy & Immunology, Omaha, Nebraska, United States